CLINICAL TRIAL: NCT04907708
Title: Comparative Studies of Metformin and Insulin on Stereological Studies and Immunohistochemistry of Placenta
Brief Title: Comparative Effects of Metformin and Insulin on Stereological Studies and Immunohistochemistry of Placenta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Responsible Party: Principal Investigator, Dr Rabia Arshad, Principal Investigator, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UKarachi
Record Dates: First submitted 2021-05-17; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Diabetes Mellitus Arising in Pregnancy, Insulin-Requiring; Diabetes Mellitus in Pregnancy
Keywords: placenta; metformin; insulin; stereology; immunohistochemistry; morphometry
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance | interventions — Metformin; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal healthy controls (No Intervention): females in second trimester with normal glucose levels
- Diet controlled (No Intervention): females in second trimester with blood sugar levels below 129mg/dl
- Metformin (Experimental): females in second trimester with blood sugar levels above 130mg/dl treated with Metformin
  Interventions: Drug: Metformin
- Insulin (Experimental): females in second trimester with blood sugar levels above 130mg/dl being treated with Insulin
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Metformin — Euglycemic agent
  Arms: Metformin
Drug: Insulin — Hypoglycemic agent
  Arms: Insulin

SUMMARY:
Diabetes mellitus is a group of metabolic disorder characterized by high blood glucose level mainly due to defect in insulin secretion or resistance. In pregnancy, insulin resistance increases as the pregnancy advances, due to the placental hormones predisposing the female to gestational diabetes mellitus (GDM). Placenta is a vital organ as it provides nutrition to the fetus. It shows morphological changes in patients with GDM leading to feto-maternal complications. Insulin, a traditional treatment given for GDM is also known to cause intra uterine deaths, stillbirths and hypoglycemia in mothers and newborns. Insulin being anabolic hormone makes placenta larger in size and causes hypoxic changes with vascular insufficiency, infarctions and hemorrhages. In contrast to this, oral insulin sensitizing drug Metformin, is euglycemic in nature. It has been proven now that Metformin is a vasculo-protective agent, with better patient compliance and beneficial micro-vascular effects in type 2 diabetics. This study was designed to clearly visualize in detail if there are any unrevealed beneficial vascular effects of Metformin on placental tissues and also to compare these effects with Insulin and diet restriction therapy, by doing placental light microscopy, morphometric studies and immunohistochemistry.

DETAILED DESCRIPTION:
Diabetes mellitus is a group of metabolic disorder with relative or absolute deficiency of insulin. Pregnancy is a potentially glucose intolerant condition as insulin sensitivity decreases with the progress of pregnancy leading to the development of gestational diabetes mellitus (GDM). It is diagnosed in approximately 3-9% of pregnancies and is growing in prevalence. In Pakistan the recent prevalence of GDM is reported to be 3-3.45% but the complications are much higher due to poor glycemic control, lack of awareness and inadequate medical facilities. Placenta is an important feto-maternal organ which is responsible for nutrition of the fetus. It also provides the retrospective information regarding infant's prenatal development. Structurally, human placenta is a complex vascular organ that allows exchange of nutrients and chemicals between fetal and maternal blood. Proper development and maturity of placenta are strongly connected with fetal growth and survival.

GDM produces anatomical and physiological alterations in placenta. This can be related to altered levels of fetal insulin and multiple growth factors such as placental vascular endothelial growth factor (VEGF), Insulin like growth factors (IGF and IGF binding proteins) which regulate the fetal and placental development. Morphologically, diabetic placentae are larger in size and volume. Microscopically, diabetic placenta shows degenerative alternations such as villous fibrinoid necrosis, chorangiosis, villous immaturity, calcification and syncytial knots formation which show intense hypoxia of the placental tissues.

Nutritional therapy (diet control) is foremost important for achieving target glucose values during pregnancy but in uncontrolled cases pharmacological intervention is required. Parental Insulin is the traditional therapy in such circumstances, but is an expensive medication and is associated with high incidence of neonatal and maternal hypoglycemia, still births, neonatal morbidity and mortality. It is documented to produce many placental alterations such as immature villi, hemorrhages, edema, cystic changes and fibrinoid necrosis. It has been postulated that the reason behind all these hypoxic changes are the variation in the blood glucose level that occur in the maternal blood as sugar level suddenly dropped soon after Insulin injection and are at highest just before the next dose of Insulin.

The use of oral anti-diabetic medications such as Metformin in the management of gestational diabetes has increased over the past several years. Recent studies has established that Metformin can be a better option for GDM as it well controls glycemia (produces euglycemic) with good pregnancy outcomes. Metformin is an oral anti-diabetic drug from biguanide group; work by improving insulin sensitivity, reducing hepatic gluconeogenesis and also by increasing peripheral glucose uptake and utilization. It is now been upgraded to category B drug as is not associated with teratogenic effects. But what are the effects of Metformin on stereological morphometric study and immunochemistry of placental tissues were left to be evaluated. Stereology provides practical measurements and significant approach for obtaining quantitative estimates of small structures on histological slides. In placental tissue it is performed to obtain unbiased quantitative estimates of placental components that inform about development and also estimate of structural parameters that have direct influence on placental functional capacity. Immunohistochemistry or immunofluorescence of tissue sections also provide valuable insight to placental structure and protein expression with three-dimensional spatial information, including morphology that cannot be obtained on microscopy.

With this background knowledge, study was designed with the following objectives:

1. To evaluate the placental gross and microscopic changes in normal, diet control, Metformin and Insulin treated in newly enrolled GDM females
2. To evaluate stereological morphometric details of placenta in normal, diet control, Metformin and Insulin all enrolled females
3. To evaluate immunohistochemistry of placental tissues in normal, diet control, Metformin and Insulin in all enrolled females
4. To compare the placental morphology, stereology and immunohistochemistry with in the groups.
5. To evaluate the fetal and maternal outcome in normal, diet control, Metformin and Insulin treated gestational diabetics.
6. To correlate the placental morphology with the fetal and maternal outcome in Metformin and Insulin treated gestational diabetics

ELIGIBILITY:
Inclusion Criteria:

For this study placentae were collected from:

1. Patients who were diagnosed as GDM during second trimester screening for FBS and RBS, confirmed further by OGCT and OGTT.
2. GDM patients who signed the written informed consent.
3. GDM patients who were in ages between 18 years and 40 years and had no other comorbid such hypertension, CVD etc
4. Full term GDM patients with singleton pregnancy (37 weeks and above)
5. GDM patients whose placenta were preserved within 30-40 minutes of delivery.

Exclusion Criteria:

Placentae were not collected from:

1. GDM Patients with ages less than 18 or more than 40 years
2. GDM females with some co-morbid and complications (e.g. hypertension, CVD, diabetes type 1 or diabetes type 2 before gestation, abnormal Urea Creatinine Electrolyte (UCE) and Liver function test (LFTs).
3. GDM Patients who delivered pre-termed (< 37 weeks of gestation) or post termed (>42 weeks of gestation)
4. GDM patients with twin pregnancy.
5. GDM Patients if not preserved in the formalin properly within 30-40 minutes of delivery.
6. GDM females who were given combined (Metformin and insulin) therapy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — GDM diagnosed pregnant females
Enrollment: 156 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Mean morphometric diffusion capacity for oxygen (MMDC) in placental tissues | 15 months
  With detailed stereological assessment MMDC can be calculated for the placenta to visualize which group placenta allows better diffusion of oxygen

SECONDARY OUTCOMES:
Percentage of immuno-antigens present in placental tissue | 15 months
  The percentage of immuno-antigens on the placental tissue is related to the hypoxic and vascular changes in the placenta.

CONTACTS AND LOCATIONS:
Overall Officials: KAUSER AAMIR, Ph.D, Study Director — BMSI, JPMC,KARACHI
Locations (1):
- Jinnah Post Graduate Medical Centre, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liang HL, Ma SJ, Xiao YN, Tan HZ. Comparative efficacy and safety of oral antidiabetic drugs and insulin in treating gestational diabetes mellitus: An updated PRISMA-compliant network meta-analysis. Medicine (Baltimore). 2017 Sep;96(38):e7939. doi: 10.1097/MD.0000000000007939. PMID 28930827
- See also: Belkacemi, L., Kjos, S., Nelson, D. M., & Desai, M. (2013). Reduced apoptosis in term placentas from gestational diabetic pregnancies. Journal of Developmental Origins of Health and Disease, 4 (3), 256-265. — https://doi.org/10.1017/S2040174413000068
- See also: Casson, I. F., Clarke, C, A., Howard, C.V., McKendrick, O., Pennycook, S., Pharoah, P.O.D. (1997). Outcomes of pregnancy in insulin dependent diabetic women: results of a five-year population cohort study, British Medical Journal, 315, 275. — http://doi.org/10.1136/bmj.315.7103.275